CLINICAL TRIAL: NCT03041987
Title: Chinese Cohort Study of Chronic Kidney Disease
Acronym: C-STRIDE
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Dongzhimen Hospital, Beijing (Other); Beijing Hospital (Other Government); Beijing Boai Hospital (Other); Peking University Shenzhen Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Guizhou Provincial People's Hospital (Other); First Affiliated Hospital of Chengdu Medical College (Other); Affiliated Hospital of Hebei University (Other); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); the Affiliated Hospital of Hubei Traditional Chinese Medical College (Unknown); Xiangya Hospital of Central South University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Chifeng Second Hospital (Unknown); The First Affiliated Hospital of BaoTou Medical College (Other); Qilu Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Second Hospital of Shanxi Medical University (Other); Minhang Central Hospital (Unknown); West China Hospital (Other); Sichuan Provincial People's Hospital (Other); Tianjin Medical University General Hospital (Other); Tianjin Medical University Second Hospital (Other); the First Affiliated Hospital of the Medical College of Shihezi University (Unknown); First Affiliated Hospital of Xinjiang Medical University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); Yuxi City People's Hospital (Unknown); Zhejiang University (Other); Xinqiao Hospital of Chongqing (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Second Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); General Hospital of Ningxia Medical University (Other); Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Minghui Zhao, Director of Renal Division, Department of Medicine, Peking University First Hospital
Other Study IDs: 2011BAI10B01
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Cohort studies; Prognosis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Urine samples DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic Kidney Disease: Specified estimated glomerular filtration rate (eGFR) range according to different CKD etiologies. For glomerular nephrology patients, the eGFR should be ≥15 ml/minute per 1.73m(2). For diabetic nephrology patients, the defining eligibility was 15 ml/minute per 1.73m(2)≤eGFR <60 ml/minute per 1.73m(2) or eGFR≥ 60 ml/minute per 1.73m(2) with "nephrotic range" proteinuria, which is defined as 24-hour urinary protein ≥3.5 g or urinary albumin creatinine ratio ≥2 000 mg/g or corresponding values of urine dipstick test or urinary protein creatinine ratio. For non-glomerular nephrology and non-diabetic nephrology patients, 15 ml/minute per 1.73m(2) ≤eGFR<60 ml/minute per 1.73m(2) is set for enrollment.
  Interventions: Other: Demographic factors, biomedical measurements, drugs used for controlling metabolic disorders, etc

INTERVENTIONS:
Other: Demographic factors, biomedical measurements, drugs used for controlling metabolic disorders, etc

SUMMARY:
This study aimed to explore underlying mechanisms of chronic kidney disease progression and its association with adverse consequences. It will enroll approximately 5000 pre-dialysis chronic kidney disease patients aged between 18 and 74 years in mainland China and follow-up for at least 5 years. Questionnaires, anthropometric measures, laboratory tests, and biomaterials will be collected at baseline and annually. The principal clinical outcomes of the study consist of renal disease events, cardiovascular events, and death.

DETAILED DESCRIPTION:
The study is a multicenter prospective cohort study, aimed to explore underlying mechanisms of chronic kidney disease progression and its association with adverse consequences. The study will establish a baseline cohort of 5000 Chinese pre-dialysis chronic kidney disease patients, who will be followed up until death or dropout or starting renal replacement therapy. The follow-up will be conducted for at least 5 years. Their clinical information and biomaterials will be collected at baseline and then annually during follow-up.

The baseline visit includes the following items: detailed demographics; socioeconomic and health care services information; medical and family history; medication history; and questionnaires concerning quality of life, health behaviors, depressive and anxiety symptoms, cognitive function, and physical activity. Anthropometric measures (height, weight, waist circumference, hip circumference, resting blood pressure, heart rate, grip strength, and 15-feet measured walk) will also be collected. The laboratory parameters of chemistry test, intact parathyroid hormone, 24-hour urine electrolytes, protein creatinine ratio, and albumin creatinine ratio should also be collected for each participant and measured in the central laboratory. After the baseline visit, participants will return annually for follow-up visits and evaluation. The evaluating items of follow-up visits are similar to the baseline visit, and sample collection.

The principal clinical outcomes of the study can be broadly categorized as renal disease events, cardiovascular events, and death. Renal disease events include the incident end stage renal disease or significant loss of renal function.Cardiovascular events include acute myocardial infarction, unstable angina, hospitalization for congestive heart failure, incident serious cardiac arrhythmia, cerebrovascular events, and peripheral vascular diseases. Death is further clarified as cardiac, cerebrovascular, renal, others, or unknown.

ELIGIBILITY:
Inclusion Criteria:

Participants should meet the following criteria of enrollment according to their etiology of nephrology.

* For glomerular nephrology patients, the estimated glomerular filtration rate (eGFR) should be ≥15 ml/minute per 1.73m(2).
* For diabetic nephrology patients, the defining eligibility was 15 ml/minute per 1.73m(2) ≤eGFR<60 ml/minute per 1.73m(2) or eGFR≥ 60 ml/minute per 1.73m(2) with "nephrotic range" proteinuria, which is defined as 24-hour urinary protein ≥3.5 g or urinary albumin creatinine ratio (ACR) ≥2 000 mg/g or corresponding values of urine dipstick test or urinary protein creatinine ratio (PCR).
* For non-glomerular nephrology and non-diabetic nephrology patients, 15 ml/minute per 1.73m(2)≤eGFR<60 ml/minute per 1.73m(2) is set for enrollment.

Exclusion Criteria:

Participants meeting even one of the listed items should be excluded.

* NYHA Class III or IV heart failure.
* Chronic kidney disease caused by systemic inflammatory illness or autoimmune disease, such as lupus erythematosus.
* Treated with immunosuppressive agents in the preceding 6 months to treat renal or immune disease.
* Self-reported or known diagnosis of HIV infection and/or AIDS.
* Isolated hematuria.
* Self-reported or known diagnosis of cirrhosis.
* Pregnant or breast-feeding women.
* Malignancy treated with chemotherapy within last 2 years.
* Renal or other transplantation.
* Hereditary kidney disease.
* Participation in interventional clinical trial.

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study enrolled chronic kidney disease patients with a broad spectrum of renal diseases with various severities and phenotypes.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
End stage renal disease or significant loss of renal function | from date of baseline examination until the date of first documented end stage renal disease or significant loss of renal function or date of death from any cause, whichever came first, up to 60 months
  start of chronic dialysis or renal transplantation or irreversible development of glomerular filtration rate <15 ml/minute per 1.73m(2) or halving of estimated glomerular filtration rate or doubling of serum creatinine compared with the value of study entry
Cardiovascular events | from date of baseline examination until the date of first documented cardiovascular events or date of death from any cause, whichever came first, up to 60 months
  acute myocardial infarction, unstable angina, hospitalization for congestive heart failure, incident serious cardiac arrhythmia (resuscitated cardiac arrest, ventricular fibrillation, sustained ventricular tachycardia, paroxysmal ventricular tachycardia, an initial episode of atrial fibrillation or flutter, severe bradycardia or heart block), cerebrovascular events (intraparenchymal hemorrhage, subarachnoid hemorrhage, cerebral infarction, cardioembolic cerebral infarction, etc.), and peripheral vascular diseases.
Death | from date of baseline examination until the date of death from any cause, up to 60 months
  death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhao, MD, Ph.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gao B, Zhang L, Wang H, Zhao M. Chinese cohort study of chronic kidney disease: design and methods. Chin Med J (Engl). 2014;127(11):2180-5. PMID 24902678
- [Result] Zhou C, Wang F, Wang JW, Zhang LX, Zhao MH. Mineral and Bone Disorder and Its Association with Cardiovascular Parameters in Chinese Patients with Chronic Kidney Disease. Chin Med J (Engl). 2016 Oct 5;129(19):2275-80. doi: 10.4103/0366-6999.190678. PMID 27647184
- [Result] Yuan J, Zou XR, Han SP, Cheng H, Wang L, Wang JW, Zhang LX, Zhao MH, Wang XQ; C-STRIDE study group. Prevalence and risk factors for cardiovascular disease among chronic kidney disease patients: results from the Chinese cohort study of chronic kidney disease (C-STRIDE). BMC Nephrol. 2017 Jan 14;18(1):23. doi: 10.1186/s12882-017-0441-9. PMID 28088175
- [Result] Peng Z, Wang J, Yuan Q, Xiao X, Xu H, Xie Y, Wang W, Huang L, Zhong Y, Ao X, Zhang L, Zhao M, Tao L, Zhou Q; C-STRIDE study group. Clinical features and CKD-related quality of life in patients with CKD G3a and CKD G3b in China: results from the Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). BMC Nephrol. 2017 Oct 13;18(1):311. doi: 10.1186/s12882-017-0725-0. PMID 29029600
- [Result] Yan Z, Wang Y, Li S, Wang J, Zhang L, Tan H, Li S, Yang L, Pei H, Zhang L, Wang Y, Duan J, Jiao S, Zhao M, Fu S; China National Survey of Chronic Kidney Disease Working Group. Hypertension Control in Adults With CKD in China: Baseline Results From the Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). Am J Hypertens. 2018 Mar 10;31(4):486-494. doi: 10.1093/ajh/hpx222. PMID 29304216
- [Result] Zhang JJ, Yang L, Huang JW, Liu YJ, Wang JW, Zhang LX, Zhao MH, Liu ZS. Characteristics and comparison between diabetes mellitus and non-diabetes mellitus among chronic kidney disease patients: A cross-sectional study of the Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). Oncotarget. 2017 Nov 10;8(63):106324-106332. doi: 10.18632/oncotarget.22368. eCollection 2017 Dec 5. PMID 29290951
- [Result] Lv L, Wang F, Wu L, Wang JW, Cui Z, Hayek SS, Wei C, Reiser J, He K, Zhang L, Chen M, Zhao MH. Soluble urokinase-type plasminogen activator receptor and incident end-stage renal disease in Chinese patients with chronic kidney disease. Nephrol Dial Transplant. 2020 Mar 1;35(3):465-470. doi: 10.1093/ndt/gfy265. PMID 30124995
- [Result] Lv L, Wang J, Gao B, Wu L, Wang F, Cui Z, He K, Zhang L, Chen M, Zhao MH. Serum uromodulin and progression of kidney disease in patients with chronic kidney disease. J Transl Med. 2018 Nov 19;16(1):316. doi: 10.1186/s12967-018-1693-2. PMID 30454063
- [Result] Yuan Q, Wang J, Peng Z, Zhou Q, Xiao X, Xie Y, Wang W, Huang L, Tang W, Sun D, Zhang L, Wang F, Zhao MH, Tao L, He K, Xu H; C-STRIDE study group. Neutrophil-to-lymphocyte ratio and incident end-stage renal disease in Chinese patients with chronic kidney disease: results from the Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). J Transl Med. 2019 Mar 15;17(1):86. doi: 10.1186/s12967-019-1808-4. PMID 30876475
- [Result] Wu L, Li XQ, Chang DY, Zhang H, Li JJ, Wu SL, Zhang LX, Chen M, Zhao MH. Associations of urinary epidermal growth factor and monocyte chemotactic protein-1 with kidney involvement in patients with diabetic kidney disease. Nephrol Dial Transplant. 2020 Feb 1;35(2):291-297. doi: 10.1093/ndt/gfy314. PMID 30357416
- [Result] Liu B, Wang Q, Wang Y, Wang J, Zhang L, Zhao M; C-STRIDE study group. Utilization of antihypertensive drugs among chronic kidney disease patients: Results from the Chinese cohort study of chronic kidney disease (C-STRIDE). J Clin Hypertens (Greenwich). 2020 Jan;22(1):57-64. doi: 10.1111/jch.13761. Epub 2019 Dec 9. PMID 31816171
- [Result] Pu L, Zou Y, Wu SK, Wang F, Zhang Y, Li GS, Wang JW, Zhang LX, Zhao MH, Wang L; C-STRIDE study group. Prevalence and associated factors of depressive symptoms among chronic kidney disease patients in China: Results from the Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). J Psychosom Res. 2020 Jan;128:109869. doi: 10.1016/j.jpsychores.2019.109869. Epub 2019 Nov 13. PMID 31739085
- [Result] Chen L, Wang J, Huang X, Wang F, Liang W, He Y, Liao Y, Zhang L, Zhao M, Xiong Z; C-STRIDE study group. Association between diabetes mellitus and health-related quality of life among patients with chronic kidney disease: results from the Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). Health Qual Life Outcomes. 2020 Aug 3;18(1):266. doi: 10.1186/s12955-020-01519-5. PMID 32746855
- [Result] Wang Q, Wang Y, Wang J, Zhang L, Zhao MH; Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). White-coat hypertension and incident end-stage renal disease in patients with non-dialysis chronic kidney disease: results from the C-STRIDE Study. J Transl Med. 2020 Jun 15;18(1):238. doi: 10.1186/s12967-020-02413-w. PMID 32539728
- [Result] Wang Q, Wang Y, Wang J, Zhang L, Zhao MH; C-STRIDE (Chinese Cohort Study of Chronic Kidney Disease)* dagger. Short-Term Systolic Blood Pressure Variability and Kidney Disease Progression in Patients With Chronic Kidney Disease: Results From C-STRIDE. J Am Heart Assoc. 2020 Jun 16;9(12):e015359. doi: 10.1161/JAHA.120.015359. Epub 2020 Jun 6. PMID 32508195
- [Result] Wang Q, Wang Y, Wang J, Zhang L, Zhao MH; Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE); Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE) Collaborators. Nocturnal Systolic Hypertension and Adverse Prognosis in Patients with CKD. Clin J Am Soc Nephrol. 2021 Mar 8;16(3):356-364. doi: 10.2215/CJN.14420920. Epub 2021 Feb 10. PMID 33568382
- [Result] Yuan Q, Xie Y, Peng Z, Wang J, Zhou Q, Xiao X, Wang W, Huang L, Tang W, Li X, Zhang L, Wang F, Zhao MH, Tao L, He K, Wanggou S, Xu H; C-STRIDE study group. Urinary magnesium predicts risk of cardiovascular disease in Chronic Kidney Disease stage 1-4 patients. Clin Nutr. 2021 Apr;40(4):2394-2400. doi: 10.1016/j.clnu.2020.10.036. Epub 2020 Oct 23. PMID 33160701
- [Result] Shen Y, Wang J, Yuan J, Yang L, Yu F, Wang X, Zhao MH, Zhang L, Zha Y; Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). Anemia among Chinese patients with chronic kidney disease and its association with quality of life - results from the Chinese cohort study of chronic kidney disease (C-STRIDE). BMC Nephrol. 2021 Feb 22;22(1):64. doi: 10.1186/s12882-021-02247-8. PMID 33618679
- [Result] Wang J, Liu L, He K, Gao B, Wang F, Zhao M, Zhang L, On Behalf Of The Chinese Cohort Study Of Chronic Kidney Disease C-Stride. UMOD Polymorphisms Associated with Kidney Function, Serum Uromodulin and Risk of Mortality among Patients with Chronic Kidney Disease, Results from the C-STRIDE Study. Genes (Basel). 2021 Oct 23;12(11):1687. doi: 10.3390/genes12111687. PMID 34828293
- [Result] Wang J, Lv J, He K, Wang F, Gao B, Zhao MH, Zhang L. Longitudinal Follow-Up and Outcomes for Chinese Patients with Stage 1-4 Chronic Kidney Disease. Kidney Dis (Basel). 2021 Oct 27;8(1):72-81. doi: 10.1159/000519190. eCollection 2022 Jan. PMID 35224008
- [Result] Wang J, Lv J, He K, Wang F, Gao B, Zhao MH, Zhang L; Chinese Cohort Study of Chronic Kidney Disease (C-STRIDE). Association of left ventricular hypertrophy and functional impairment with cardiovascular outcomes and mortality among patients with chronic kidney disease, results from the C-STRIDE study. Nephrology (Carlton). 2022 Apr;27(4):327-336. doi: 10.1111/nep.14009. Epub 2021 Dec 15. PMID 34843156
- [Result] Deng X, Gao B, Wang F, Zhao MH, Wang J, Zhang L. Red Blood Cell Distribution Width Is Associated With Adverse Kidney Outcomes in Patients With Chronic Kidney Disease. Front Med (Lausanne). 2022 Jun 9;9:877220. doi: 10.3389/fmed.2022.877220. eCollection 2022. PMID 35755057
- [Result] Hui M, Ma J, Yang H, Gao B, Wang F, Wang J, Lv J, Zhang L, Yang L, Zhao M. ESKD Risk Prediction Model in a Multicenter Chronic Kidney Disease Cohort in China: A Derivation, Validation, and Comparison Study. J Clin Med. 2023 Feb 14;12(4):1504. doi: 10.3390/jcm12041504. PMID 36836039
- [Result] Xue X, Li JX, Wang JW, Lin LM, Cheng H, Deng DF, Xu WC, Zhao Y, Zou XR, Yuan J, Zhang LX, Zhao MH, Wang XQ. Association between alkaline phosphatase/albumin ratio and the prognosis in patients with chronic kidney disease stages 1-4: results from a C-STRIDE prospective cohort study. Front Med (Lausanne). 2023 Sep 20;10:1215318. doi: 10.3389/fmed.2023.1215318. eCollection 2023. PMID 37799589